CLINICAL TRIAL: NCT02323542
Title: Plasma Glucose Kinetics Following Ingestion of Two Cereal Products With a Different Content in Slowly Digestible Starch (SDS) in Healthy Males and Females
Brief Title: Plasma Glucose Kinetics and Cereal Product Content in Slowly Digestible Starch (SDS) in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: Institut de Recherches Cliniques de Montreal (Other); Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other); BioFortis (Other); MedQualis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KBE032
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Blood Glucose Kinetics
Keywords: Starch; cereal products; glucose kinetics; blood glucose; blood insulin
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-SDS biscuit (Experimental): Biscuit with high Slowly Digestible Starch content
  Interventions: Other: Nutrition intervention with cereal products
- Low-SDS cereal product (Active Comparator): Cereal product with low Slowly Digestible Starch content
  Interventions: Other: Nutrition intervention with cereal products

INTERVENTIONS:
Other: Nutrition intervention with cereal products — acute evaluation of the effect of ingestion of cereal products differing by their Slowly Digestible Starch content

SUMMARY:
The present study aims at investigating the effect of ingesting 2 cereal products differing by their SDS content on the kinetics of glucose in healthy volunteers.

DETAILED DESCRIPTION:
The present study will compare the effect of consuming cereal products alone on :

* the rates of appearance and disappearance of exogenous and total glucose
* the glycemic and insulinemic responses
* the postprandial GIP concentrations

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer, male or female (half male, half female);
* Aged between 18 and 40 years old (bounds included);
* Non-smoker;
* BMI ranging between 18.5 and 25 kg/m2 (bounds included)
* Waist circumference ≤ 94 cm for men and ≤ 80 cm for women;
* Stable body weight (± 1 kg) over the 3 months preceding the experimental period;
* Systolic blood pressure between 95 and 145 mmHg and diastolic blood pressure between 50 and 85 mmHg;
* For the female subjects: use of an oral contraceptive with regular menstrual cycles;
* Subject not displaying any identified significant metabolic impairment according to the Principal Investigator;
* Sedentary or with a moderate physical activity;
* Not having given blood in the month prior to the selection and accepting not to give blood during the experimental period of the present study;
* Regularly consuming a breakfast providing more than 15% of the total daily energy intake, including at least one cereal product; adequate partitioning of macronutrient intake;
* Providing written consent for his/her participation to the study;

Exclusion Criteria:

* Subject with a severe or acute disease which should influence the results of the study and to be life-threatening for the volunteer according to the Principal Investigator;
* Subject with medical history of symptomatic vascular diseases (infarct, angina pectoris, syndrome of threat, surgery or endovascular surgery, stroke, symptomatic peripheral arteritis) which according to the investigator should interfere with the results from the study or should constitute a particular risk for the subject;
* Subject with type 1 or type 2 diabetes;
* Subject with any food allergy;
* Subject with eating disorders (e.g. anorexia nervosa & bulimia) according to the Principal Investigator;
* Subject regularly consuming more than 20 g/day of alcohol;
* Subject regularly consuming recreational drugs;
* Subject consuming regularly corticoids, anorectics, adrenergic drugs, gastric demulcent, cholesterol and/or lipid lowering medication, weight-loss drugs or other drugs or supplement that should impact glucose metabolism in the Principal Investigator's opinion;
* Pregnant or lactating women;
* Currently participating in another study or having participated in another study in the 3 months prior to the selection visit;
* Consuming large amounts of food products naturally rich in 13C.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Rate of appearance of exogenous glucose (RaE) | T0 to 300 minutes
  Postprandial kinetic of RaE

SECONDARY OUTCOMES:
iAUC RaE | T0 to 300 minutes
  iAUC of RaE over selected intervals over the 300-minute postprandial period
kinetics of Rate of disappearance of exogenous glucose (RdE), Rate of appearance of total glucose (RaT), Rate of disappearance of total glucose (RdT) and Endogenous glucose production (EGP) | T0 to 300 minutes
  Postprandial kinetics of RdE, RaT, RdT and EGP
iAUC of RdE, RaT, RdT and EGP | T0 to 300 minutes
  iAUC of RdE, RaT and RdT and dAUC of EGP over selected intervals over the 300-minute postprandial period
kinetics of glycemia and insulinemia | T-120 to 300 minutes
  Pre- and postprandial kinetics of glycemia and insulinemia
iAUC of glycemia and insulinemia | T0 to 300 minutes
  iAUC of glycemia and insulinemia over selected intervals over the 300-minute postprandial period
Kinetics of plasma glucose-dependent insulinotropic peptide (GIP) concentration | T0 to 300 minutes
  Postprandial kinetic of GIP
iAUC of GIP | T0 to 300 minutes
  iAUC of GIP over selected intervals over the 300-minute postprandial period
Kinetics of plasma FFA concentration | T0 to 300 minutes
  Postprandial kinetic of FFA
dAUC of FFA | T0 to 300 minutes
  dAUC of FFA over selected intervals over the 300-minute postprandial period

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Llhoret, MD, PhD, Principal Investigator — Institut de Recherches Cliniques de Montreal
Locations (1):
- Institut de Recherches Cliniques de Montréal, Montreal, Quebec, Canada